CLINICAL TRIAL: NCT02234869
Title: Open-label, Randomized, 2-arm, Active Comparator Study to Evaluate Safety and Tolerability in Patients With Relapsing Multiple Sclerosis Transitioning From Standard-of-care Subcutaneous Interferon Therapy to Peginterferon Beta-1a (BIIB017)
Brief Title: Transition to Peginterferon Beta-1a (BIIB017) From Subcutaneous Interferon Therapy
Acronym: Frequency
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to a change in Biogen Idec's medical research plans.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105MS403
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Peginterferon Beta-1a; Relapsing Multiple Sclerosis; RMS; flu-like symptoms
MeSH Terms: interventions — Interferon-beta; Interferon beta-1a; Interferon beta-1b; peginterferon beta-1a

ARMS (2):
- Peginterferon beta-1a (Experimental): Participants will receive peginterferon beta-1a, 125 µg subcutaneously once every 2 weeks during the 6-month comparator period of the study and during the 12-month extension period.
  Interventions: Drug: BIIB017 (Peginterferon beta-1a)
- Interferon-β (Active Comparator): Participants will continue to receive their standard-of-care interferon beta treatment for the first six months. During the 12-month extension period participants will switch to receive peginterferon beta-1a, 125 µg subcutaneously once every 2 weeks.
  Interventions: Drug: Interferon Beta; Drug: BIIB017 (Peginterferon beta-1a)

INTERVENTIONS:
Drug: Interferon Beta — Subcutaneous injection
  Other Names: Rebif or Betaseron/Betaferon
  Arms: Interferon-β
Drug: BIIB017 (Peginterferon beta-1a) — Single-use, disposable, prefilled pen for subcutaneous injection
  Other Names: PEGylated interferon beta-1a (IFN β-1a)

SUMMARY:
The primary objective of the study is to evaluate, in participants with RMS, safety and tolerability (as defined by the frequency of adverse events [AEs] of flu-like symptoms [FLS; chills, pyrexia, myalgia, and asthenia], injection site reactions [ISRs], and injection site reaction pain [ISR-P]) over 6 months of treatment (the active comparator period) with BIIB017 125 μg subcutaneously (SC) every 2 weeks versus standard-of-care SC interferon-beta (IFN-β) therapy. Secondary objectives of this study are to assess the following measures during the first (6-month) period of the study in participants treated with BIIB017 versus standard-of-care SC IFN-β therapy: patient-reported treatment satisfaction using the following patient-reported outcome measures (PROMs): Treatment Satisfaction Questionnaire for Medication (TSQM-9), Adapted MS Treatment Concerns Questionnaire (MSTCQ), Adapted MSTCQ Side Effects Score, Pain using a visual analog scale (VAS) diary and the McGill Pain Questionnaire Short Form (SF-MPQ), the treatments' impact on RMS using the following PROMs: Multiple Sclerosis Impact Scale (MSIS-29), Modified Fatigue Impact Scale-5 Item (MFIS-5), EuroQol Group 5-Dimension 3-Level Version (EQ-5D-3L), Health-Related Productivity Questionnaire (HRPQ), Beck Depression Inventory, second edition (BDI-II), participant adherence to study treatment, clinical status as measured by the Expanded Disability Status Scale (EDSS) and relapse activity, safety and tolerability of study treatment after a change in standard-of-care SC IFN-β therapy and the immunogenicity profiles of participants changing from standard-of-care SC IFN-β to BIIB017.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a confirmed diagnosis of Relapsing Multiple Sclerosis (RMS), as defined by McDonald criteria.
* An Expanded Disability Status Scale (EDSS) score between 0 and 5.0.
* On continual treatment for ≥6 months with a single standard-of-care subcutaneous (SC) interferon beta (IFN-β) therapy, including IFN β-1b 0.25 mg SC every other day or IFN β-1a 44 μg SC 3 times weekly, and from a clinical perspective be able to continue this therapy (i.e., no significant untoward events attributed to IFN therapy that would preclude continuation of the existing IFN therapy).
* A candidate for change to BIIB017 therapy (candidacy for therapy change is determined by the treating physician; however, it is recommended to exclude patients with high disease activity and who are candidates for escalation therapy according to local guidelines).
* Patients who are randomized to their current standard-of-care IFN-β therapy for the first 6 months of the study must be willing to receive their treatment via the formulation provided in the study (i.e., Rebif 44 μg in a prefilled syringe or Betaferon/Betaseron 0.25 mg in single-use vials of lyophilized powder accompanied by a prefilled single-use diluent syringe).

Key Exclusion Criteria:

* Primary progressive, secondary progressive, or progressive relapsing MS.
* History of inadequate response to SC IFN therapy (as determined by the treating physician).
* History of severe allergic or anaphylactic reactions or known hypersensitivity to study drug or its excipients. - Known allergy to any component of the BIIB017 formulation.
* History of any clinically significant (as determined by the Investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease that would preclude participation in a clinical study.
* History of hypersensitivity or intolerance to acetaminophen, ibuprofen, naproxen, or aspirin that would preclude use of at least one of these during the study.
* An MS relapse that has occurred within the 50 days prior to randomization and/or lack of stabilization from a previous relapse prior to randomization.
* Any previous treatment with BIIB017.
* Treatment with other agents for MS.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2017-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Combined Counts of adverse events (AEs) of flu-like symptoms, injection site reactions or injection site reaction pain | 6 Months
  Combined counts of AEs of flu-like symptoms (FLS) including chills, pyrexia, myalgia, and asthenia, injection site reactions (ISRs), and injection site reaction pain (ISR-P) over the first 6 months of treatment.

SECONDARY OUTCOMES:
Change from Baseline in treatment satisfaction using the Treatment Satisfaction Questionnaire for Medication-9 Items (TSQM-9) | Baseline and Week 24
  The TSQM-9 is a 9-item, validated questionnaire that assesses participants' satisfaction with treatment and captures information on treatment effectiveness, convenience, and overall satisfaction.
Change from Baseline in adapted Multiple Sclerosis Treatment Concerns Questionnaire (MSTCQ) total score | Baseline and Week 24
  The adapted MSTCQ self-administered questionnaire includes evaluation of the injection process, treatment differences, overall injection issues, FLS, and ISRs.
Change from Baseline in the adapted MSTCQ Side Effects Score | Baseline and Week 24
Percentage of participants pain-free | 6 months
  Pain free is defined as a score of 0 for all full-dose injections measured on a visual analog scale (VAS) diary of patient-reported pain. The scale ranges from 0 (no pain) to 10 (worse possible pain).
Change from Baseline in mean change in VAS pain score from pre-injection to 30 minutes post-injection | Baseline (pre-injection and 30-minutes after injection) and Week 24 (pre-injection and 30 minutes after injection)
  Pain was measured on a visual analog scale (VAS) prior to injection and 30 minutes after injection. The VAS scale ranges from 0 (no pain) to 10 (worse possible pain).
Change from Baseline in mean McGill Pain Questionnaire Short Form (SF-MPQ) VAS pain score | Baseline and Week 24
  This self-administered questionnaire provides qualitative measures of clinical pain that captures its sensory, affective, and other qualitative components.
Change from Baseline in the Multiple Sclerosis Impact Scale-29 items (MSIS-29) score | Baseline and Week 24
  The MSIS-29 is a self-report questionnaire measuring the physical (20 items) and psychological (9 items) impact of MS from the patient's perspective. Each of the 29 questions can take 1 of 5 responses, ranging from 1 (not at all) to 5 (extremely). Combined scores for MSIS-29 scales are generated by summing items, with a total score ranging from 29 to 145.
Change from Baseline in the Modified Fatigue Impact Scale-5 Item (MFIS-5) score | Baseline and Week 24
  The MFIS-5 is a structured, self-report questionnaire, modified from the Fatigue Impact Scale. The abbreviated version (MFIS-5) has 5 items taken from the physical (2 items), cognitive (2 items), and psychological (1 item) subscales of the standard 21-item MFIS. The participant is asked to score each item from 0 to 4. All items are scaled so that higher scores indicate a greater impact of fatigue on a participant's activities. The MFIS-5 total score consists of the sum of the raw scores on the 5 items, and thus can range from 0 to 20.
Change from Baseline in the EuroQol-5-dimension 3-level version (EQ-5D-3L) index | Baseline and Week 24
  The EQ-5D-3L is a descriptive system of health-related quality-of-life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which can take 1 of 3 responses. The responses record 3 levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension.
Change from Baseline in the Health-Related Productivity Questionnaire (HRPQ) score | Baseline and Week 24
  This self-administered questionnaire provides information about absenteeism and presenteeism over the previous week and includes an estimate of unproductive work time.
Change from Baseline in the Beck Depression Inventory, second edition (BDI-II) score | Baseline and Week 24
  BDI-II is a 21-item self-administered questionnaire to assess the intensity of depression.
Percentage of participants with changes in Clinical Status assessed using the Expanded Disability Status Scale (EDSS) | Up to 6 months
  The EDSS is a method of quantifying disability in MS. The EDSS is an ordinal clinical rating scale based on a standard neurological exam, with scores ranging from 0 (normal neurological exam) to 10 (death due to MS) in half-point increments.
Annualized relapse rate (ARR) | 6 months
  The ARR is calculated by dividing the number of relapses the participants experience during a 1-year period by the number of participants.
Percentage of participants with relapse | 6 months
  A clinical relapse is defined as new or recurrent neurological symptoms not associated with fever or infection, lasting for at least 24 hours, and accompanied by new objective neurologic findings on examination by a neurologist.
Adherence to study treatment measured by returned autoinjectors/syringes | 6 months
Adherence to study treatment measured by the treatment adherence questionnaire | 6 months
Number of participants with adverse events (AEs), serious adverse events (SAEs), and discontinuations of study treatment due to an AE | 6 months
Number of participants with IFN β-1a and IFN β-1b binding and neutralizing antibodies, and poly(ethylene glycol) (PEG)-binding antibodies | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen